CLINICAL TRIAL: NCT01415011
Title: Trial of Afatinib (BIBW 2992) in Suspected or Confirmed Mutant EGFR Lung Cancer Patients Unfit for Chemotherapy
Brief Title: Efficacy and Safety Study of Afatinib to Treat Lung Cancer Patients
Acronym: TIMELY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/09/0426; 2011-003608-19 (EudraCT Number)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2017-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Afatinib (BIBW2992); EGFR Mutation; Non Small Cell Lung Cancer; Poor performance status; Elderly
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Afatinib (BIBW 2992) (Experimental): All patients will be given daily oral afatinib (BIBW 2992) administered every 28 days until disease progression/toxicity/clinician decision to stop. Starting dose is 40mg. 30mg and 20mg will be administered according to protocol dose modification requirements following toxicity.
  Interventions: Drug: Afatinib (BIBW 2992)

INTERVENTIONS:
Drug: Afatinib (BIBW 2992) — All patients will be given daily oral afatinib (BIBW 2992) administered every 28 days until disease progression/toxicity/clinician decision to stop. Starting dose is 40mg. 30mg and 20mg will be administered according to protocol dose modification requirements following toxicity.

SUMMARY:
The purpose of this study is to examine the efficacy and safety of using afatinib (BIBW 2992) to treat non-small cell lung cancer patients considered unfit for chemotherapy and have either suspected or confirmed Epidermal Growth Factor Receptor (EGFR) mutation.

DETAILED DESCRIPTION:
Lung cancer is most common cause of death from cancer, of which non-small cell lung cancer (NSCLC) accounts for ~80% of all cases with most patients presenting with advanced disease. Patients medically unfit to receive radical or platinum-doublet palliative systemic therapy, because of poor performance status or comorbidity, account for at least 45% of newly diagnosed cases and have poor survival. Many oncologists have interpreted single-agent chemotherapy data as not clinically meaningful when balanced against toxicities, non-significant improvements in quality of life and comorbidity. Hence, in the UK, this group of patients are predominantly treated by best-supportive care (BSC).

This study aims to examine the efficacy and safety of using afatinib (BIBW 2992), an irreversible second generation EGFR inhibitor, in patients with non-small cell lung cancer, who are considered unfit for chemotherapy and have either suspected or confirmed Epidermal Growth Factor Receptor (EGFR) mutation.

Suspected EGFR mutant patients will have clinical characteristics likely to harbour the EGFR mutation (adenocarcinoma sub type and ex or never smokers) with EGFR genotype unknown either due to no tissue suitable for genotyping or failed genotype.

There has been only one small prospective study of medically unfit patients with EGFR mutation, but it demonstrated good efficacy with a TKI17. This phase II study of East Asian patients (n=30) with performance status 2-4 and treated with gefitinib demonstrated a rapid improvement in performance status at 1 month, an overall response rate of 66% and median survival of 17.8 months. Whilst gefitinib is licensed for EGFR mutant NSCLC, no prospective studies have yet been performed on medically unfit patients from Western countries. Despite dramatic initial responses, EGFR mutant NSCLC patients treated with gefitinib/erlotinib ultimately relapse. In ~50% of cases this is due to the gefitinib/erlotinib-resistant T790M genotype acquired through either secondary somatic mutation or clonal expansion. There is therefore a need to improve the outcomes of medically unfit patients with suspected EGFR mutation, who would otherwise be treated with best supportive care, and in proven EGFR mutation cases by using an effective EGFR-directed therapy that inhibits EGFRT790M.

Prospective data on medically unfit Western NSCLC patients with EGFR mutation are required to assess the efficacy of EGFR-TKIs. Additionally, given that 50% of such patients will become TKI-resistant through EGFRT790M, new therapies are required to overcome this resistance mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Any stage not suitable for radical treatment
* Either:

Confirmed activating EGFR mutation (exons 18-21; e.g. L858R, exon 19 deletions, exon 20 insertions, T790M, list is not exhaustive), and WHO PS 0-3 Or No tissue suitable for EGFR genotyping, failed genotype, or EGFR genotyping unavailable, and NSCLC Adenocarcinoma sub-type, and

Eligible smoking history:

Never smoker (<100 cigarettes in lifetime), or Former smoker (stopped >1year ago and ≤10 pack-years) and WHO PS 0-2

* Unsuitable for or patient declining chemotherapy due to significant co-morbidity
* Measurable disease according to RECIST version 1.1
* Adequate haematopoietic, hepatic and renal function defined as follows:

Absolute neutrophil count (ANC) ≤1.5 x 109/L and platelet count ≤100 x 109/L

* Bilirubin ≤1.5 x ULN, ALT (SGPT) ≤3 x ULN (or ≤ 5 x ULN in cases of liver metastases)
* Serum creatinine clearance ≥45 ml/min
* Palliative radiotherapy allowed unless to a solitary target lesion
* Age 18 or over (no upper age limit)
* Written informed consent that is consistent with ICH-GCP guidelines

Exclusion Criteria:

* Previous treatment with afatinib (BIBW 2992), or any EGFR-directed inhibitor
* Any concurrent anticancer systemic therapy
* Prior chemotherapy for relapsed and/or metastatic NSCLC
* Neoadjuvant/adjuvant chemotherapy is permitted if at least 12 months has elapsed between the end of chemotherapy and registration
* Suitable for radical radiotherapy
* Palliative radiotherapy within 2 weeks prior to registration
* Palliative radiotherapy to a solitary target lesion
* Surgery (other than biopsy) within 4 weeks prior to registration
* Inability to take oral medication, requirement for intravenous feeding, active peptic ulcer, prior surgical procedures affecting absorption, any medical co- morbidity affecting gastrointestinal absorption
* Patients with current or pre-existing interstitial lung disease
* Active or uncontrolled infections or serious illnesses or medical conditions that could interfere with the patient's participation in the trial
* Significant or recent acute gastrointestinal abnormalities with diarrhoea as a major symptom e.g., Crohn's disease, mal-absorption, or CTCAE version 4.0 Grade ≥3 diarrhoea of any etiology at baseline
* Active brain metastases (defined as stable for <4 weeks and/or symptomatic and/or requiring treatment with anticonvulsants and/or leptomeningeal disease). Steroids will be allowed if administered as a stable (same) dose for at least one month before trial entry.
* Any other current malignancy or malignancy diagnosed within the past five years (other than non-melanomatous skin cancer and in situ cervical cancer)
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3 or more, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to registration
* Symptomatic left ventricular failure with NYHA classification of 3 or more
* Active viral hepatitis and/or known HIV positive
* Known or suspected active drug or alcohol abuse
* Use of any investigational drug within 8 weeks of registration.
* Known allergy to BIBW 2992 or other ingredients.
* Patients on steroids must have been on the same dose for at least 4 weeks.
* Inability to understand or to comply with the requirements of the trial, trial protocol or to provide informed consent.
* Women of childbearing potential, or men who are able to father a child, unwilling to use a medically acceptable method of contraception during the trial
* Women who are pregnant or breast feeding
* Requirement for treatment with any of the prohibited concomitant medications listed in protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-12; Primary Completion 2015-08 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival | At 6 months
  Progression free survival will be determined by measurement of tumour size using RECIST version 1.1 at progression or date of patient death.

SECONDARY OUTCOMES:
Overall response | CT scan of chest & abdomen 4 weeks after registartion, then every 8 calender weeks until disease progression. CT scans every 12 weeks if patient is still on BIBW 2992 after 1 year of treatment.
Overall survival | This will be measured in days, from the first day of treatment to the day of death.
Change in performance status | At 1 month
Safety | To be assessed at every timepoint i.e. baseline, fortnightly for the first 2 cycles and then monthly for 12 months and 2 monthly thereafter
  For each type of adverse event, the maximum toxicity grade will be obtained for each patient using CTCAE version 4.0 to closely monitor tolerability to BIBW 2992. Focus will be on those with a grade 3 or 4 BIBW 2992 related toxicities. The proportion of patients with any grade 3 or 4 event will also be examined.
Progression free survival in patients aged 70 and over | At progression or patient death
Treatment compliance | Compliance will be examined based on the time between starting treatment and stopping it completely

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Popat, BSc MBBS MRCP PhD, Principal Investigator — Royal Marsden Hospital London
Locations (15):
- United Kingdom (15):
  - Royal Bournemouth Hospital, Bournemouth
  - Beatson West of Scotland Cancer Centre, Glasgow
  - James Paget University Hospital, Great Yarmouth
  - East Kent Hospitals, Kent
  - Maidstone Hospital, Kent
  - St James's University Hospital, Leeds
  - Barnet & Chase Farm Hospitals, London
  - Charing Cross Hospital, London
  - Guy's Hospital, London
  - University College Hospital, London
  - Musgrove Park Hospital, Somerset
  - The Royal Marsden Hospitals, Sutton
  - King's Mill Hospital, Sutton in Ashfield
  - Weston General Hospital, Weston-super-Mare
  - York Hospital, York

REFERENCES:
- See also: Cancer Research UK & UCL Cancer Trials Centre — http://www.ctc.ucl.ac.uk